CLINICAL TRIAL: NCT04109196
Title: Examining Changes in Microbiota Over the Course of PTSD Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Chicago (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Philip Held, Research Director, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18011005; 5KL2TR002387-02 (NIH)
Record Dates: First submitted 2019-09-06; First posted 2019-09-30 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Posttraumatic Stress Disorder; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Intervention Model Description: All participants who are eligible for this study will receive a 5 day PTSD treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive 5-day Cognitive Processing Therapy for PTSD (Experimental): Participants who are eligible for and enrolled in the study will receive a 5-day CPT treatment for PTSD. All participants will be asked to complete clinician-rated and self-report assessments at multiple time points during the study. Participants will also be asked to provide fecal and saliva samples as part of the study, however, they may opt out of biological sample collection.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy is an evidence-based treatment for PTSD that will be delivered intensively twice per day over the course of five days.

SUMMARY:
The overall goals of this project are to evaluate the use of 5-day intensively-delivered Cognitive Processing Therapy to treat PTSD and to determine the associations between the microbiome, salivary cytokines, and the presence of and recovery from PTSD. Specifically, this study is designed to 1) determine whether individual Cognitive Processing Therapy (CPT) delivered twice per day over 5 consecutive days (CPT-5) is tolerable, acceptable, and effective in reducing PTSD symptoms, 2) determine the microbial signatures associated with PTSD, 3) evaluate whether the abundance and composition of microbiota and salivary cytokine levels change over the course of PTSD treatment, and 4) examine whether changes in microbial signatures are associated with changes in cytokine levels.

DETAILED DESCRIPTION:
This project will evaluate the use of 5-day intensively-delivered Cognitive Processing Therapy to treat PTSD and will aim to determine the associations between the microbiome, salivary cytokines, and the presence of and recovery from PTSD. A total of 24 participants who have experienced a criterion A trauma will be recruited. An intake assessment will be used to confirm the fit for the proposed project. Clinical interviewers with a minimum of a Master's degree in Psychology who are not providing the treatment will administer structured diagnostic interviews (CAPS and DIAMOND). If an individual meets criteria for a PTSD diagnosis based on the CAPS they will be eligible for this treatment study.

Study staff will administer brief computerized assessments (e.g. Stroop task), a full self-report assessment battery, and two internet-based dietary assessments to all participants. Study staff will also collect fecal- and oral-derived microbiota and salivary cytokine samples from individuals who opt in to this aspect of the study.

Study Treatment - Intensive Week-Long Cognitive Processing Therapy (CPT):

The individuals in this study will undergo a course of 1-week-long Cognitive Processing Therapy (CPT-5). CPT-5 will be delivered twice per day over the course of five business days. Each 50 minute session will closely follow the CPT protocol and will be conducted by either Dr. Held, other doctoral-level psychologists, postdoctoral fellows, or other Master's level (or higher) clinicians who have received the official two-day CPT training and who are not involved in study assessments. CPT worksheets and homework assignments may be collected and copied for research purposes. Changes in PTSD severity and other relevant symptoms will be assessed before, during, and after the course of CPT using well-validated clinician-administered, self-report, and computerized assessments. Fecal- and oral-derived microbiota as well as salivary cytokines will also be assessed at various pre-treatment, post-treatment, and follow-up time points to determine whether the microbiome and cytokine levels change over the course of CPT. Participants in this study will have the option to opt out of providing these biological samples and still receive CPT-5.

Semi-Structured Interview:

Regardless of whether they completed the course of CPT, participants in the study may be asked to participate in one 20-40 minute semi-structured interview. The interviewer, who is a member of the research team and not the respective participant's study therapist, will ask general questions about the participant's experiences of CPT-5 and gather information about the participant's perceptions of the tolerability, acceptability, and feasibility of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Individuals are eligible for the study if they:

1. Are 18 years or older
2. Are fluent in English
3. Have experienced a Criterion A traumatic event during their lifetime
4. Have a PTSD diagnosis verified by the Clinician Administered PTSD Scale for DSM-5
5. Are interested in receiving evidence-based treatment (CPT) for PTSD and able to attend 10 therapy sessions over the course of one week (5 days)
6. Are willing and interested to complete self-report measures and clinician-rated assessments at multiple time points over the course of the study

Exclusion Criteria:

Individuals are excluded from the study if:

1. The traumatic event occurred in the past month
2. They are currently suicidal or homicidal, as indicated by a positive screen on the C-SSRS Question 4 or Question 5 at intake.
3. They have a history of psychosis or mania
4. They have not been on a stable dose of medication for at least one month
5. They have dietary patterns not representative of normal populations (e.g., vegetarian, vegan, gluten-free)
6. They made changes to the diet in the past month or are planning to make changes over the course of therapy
7. They have completed an evidence-based PTSD treatment in the past 3 months or are currently receiving an evidence-based PTSD treatment
8. They have mental retardation or significant cognitive impairment that would prevent them from engaging in CPT
9. They have a serious or unstable medical illness or instability for which hospitalization may be likely within the next year
10. They have an active substance use disorder (within the past 3 months)
11. They are involved with current legal actions related to the traumatic event that is anticipated to be targeted during treatment
12. They have a history or presence of an eating disorder
13. They are currently taking or have taken an antibiotic in the past 30 days
14. They are currently taking a corticosteroid
15. They have had part of the digestive tract removed or altered
16. They have had any surgery or procedure within the past 30 days that has required fasting for more than 12 hours or bowel preparation beforehand
17. They are unwilling to provide fecal and saliva samples (applies to trauma-exposed control condition only)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (121.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 17
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: This will be used to assess severity of posttraumatic stress disorder symptoms at intake.The PTSD Checklist for DSM-5 (PCL-5) measures severity of PTSD symptoms. This questionnaire includes 20 items, which each item rated on a scale of 0 (not at all)-4 (extremely). There are four subscales reflecting symptom clusters in the DSM-5: intrusion (five items), avoidance (two items), negative alterations in cognitions and mood (seven items), and alterations in arousal and reactivity (six items). All 20 items are summed to calculate a total score. Scores range from 0-80, with higher scores indicating more severe symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 24
score on a scale | 53.08 (12.81)

2. Primary Outcome: Change in PTSD Checklist for DSM-5 (PCL-5) From Baseline
Description: This will be used to assess changes in posttraumatic stress disorder symptom severity from baseline to the time points described below and/or changes between the time points described below. The PTSD Checklist for DSM-5 (PCL-5) measures severity of PTSD symptoms. This questionnaire includes 20 items, which each item rated on a scale of 0 (not at all)-4 (extremely). There are four subscales reflecting symptom clusters in the DSM-5: intrusion (five items), avoidance (two items), negative alterations in cognitions and mood (seven items), and alterations in arousal and reactivity (six items). All 20 items are summed to calculate a total score. Scores range from 0-80, with higher scores indicating more severe symptoms.
Time Frame: 1 week post-treatment, 3 months post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 24
score on a scale
  1-week post-treatment | 17.55 (14.11)
  3-months post-treatment | 19.42 (15.75)

3. Primary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: This will be used to assess severity of depression symptoms at intake. The Patient Health Quetionnaire-9 (PHQ-9) measures severity of depression symptoms. This questionnaire includes 10 items, with each item rated on a scale of 0 (not at all)-3 (nearly every day). The first 9 items are summed to calculate a total score. Scores range from 0-27, with higher scores indicating more severe symptoms. The tenth item (also rated 0-3) is not included in the total score, but indicates how much interference the responder experiences in their day to day life due to symptoms they are experiencing.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 24
score on a scale | 15.38 (4.97)

4. Primary Outcome: Change in Patient Health Questionnaire-9 (PHQ-9) From Baseline
Description: This will be used to assess changes in depression symptom severity from baseline to the time points described below and/or changes between the time points described below. This will be used to assess severity of depression symptoms at intake. The Patient Health Quetionnaire-9 (PHQ-9) measures severity of depression symptoms. This questionnaire includes 10 items, with each item rated on a scale of 0 (not at all)-3 (nearly every day). The first 9 items are summed to calculate a total score. Scores range from 0-27, with higher scores indicating more severe symptoms. The tenth item (also rated 0-3) is not included in the total score, but indicates how much interference the responder experiences in their day to day life due to symptoms they are experiencing.
Time Frame: 1 week post-treatment, 3 months post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 24
score on a scale
  1-week post-treatment | 7.73 (5.51)
  3-months post-treatment | 6.84 (5.47)

5. Primary Outcome: Change in DNA Genotek OMNIgeneGUT for Microbiome Kit (OMR-200) From Baseline
Description: Change in microbial signature (abundance and composition) from colonic fecal sample from baseline to the time points described below and/or changes between the time points described below.
Time Frame: Intake, Day 1 of treatment, 1 week post-treatment, 3 months post-treatment
Population: This part of the study was discontinued as COVID protocols required the study to move to a virtual format where this type of data was unable to be collected.
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 0

6. Primary Outcome: DNA Genotek OMNIgeneORAL for Collection of Microbial DNA Kit (OM-501)
Description: Microbial signature (abundance and composition) from oral saliva sample collected at intake.
Time Frame: Baseline
Population: as for outcome 5
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 0

7. Primary Outcome: Change in DNA Genotek OMNIgeneORAL for Collection of Microbial DNA Kit (OM-501) From Baseline
Description: Change in microbial signature (abundance and composition) from oral saliva sample from baseline to the time points described below and/or changes between the time points described below.
Time Frame: Intake, Day 1 of treatment, 1 week post-treatment, 3 months post-treatment
Population: as for outcome 5
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 0

8. Primary Outcome: Salimetrics Salivary Cytokine Panel
Description: Salivary cytokine levels (TNF-alpha, IL-1beta, IL-6, IL-8) from oral saliva sample collected at intake.
Time Frame: Baseline
Population: as for outcome 5
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 0

9. Primary Outcome: Change in Salimetrics Salivary Cytokine Panel From Baseline
Description: Change in salivary cytokine levels (TNF-alpha, IL-1beta, IL-6, IL-8) from baseline to the time points described below and/or changes between the time points described below.
Time Frame: Intake, Day 1 of treatment, 1 week post-treatment, 3 months post-treatment
Population: as for outcome 5
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 0

10. Secondary Outcome: Posttraumatic Cognitions Inventory (PTCI)
Description: Will be used to assess intensity of negative posttrauma cognitions at intake. The PTCI score is calculated by summing all items, with scores ranging from 22 to 231. Higher scores indicate more severe negative cognitions.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 24
score on a scale | 154.08 (36.71)

11. Secondary Outcome: Change in Posttraumatic Cognitions Inventory (PTCI) From Baseline
Description: Will be used to assess changes in intensity of negative posttrauma cognitions from baseline to the time points described below and/or changes between the time points described below. The PTCI score is calculated by summing all items, with scores ranging from 22 to 231. Higher scores indicate more severe negative cognitions.
Time Frame: 1 week post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
Number analyzed (Participants) | 24
score on a scale | 89.23 (43.09)

ADVERSE EVENTS:
Time Frame: Data were collected from Baseline to 3 months follow up.
Arm/Group | Intensive 5-day Cognitive Processing Therapy for PTSD
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT04109196/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT04109196/SAP_001.pdf